CLINICAL TRIAL: NCT05877781
Title: THE EFFECT OF DIETARY SUPPLEMENTATION WITH PALMITOYLETHANOLAMIDE ON GASTROINTESTINAL SYMPTOMS IN FUNCTIONAL DYSPEPSIA PATIENTS.
Brief Title: PEA in Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S65406
Record Dates: First submitted 2023-03-06; First posted 2023-05-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Dyspepsia and Other Specified Disorders of Function of Stomach
MeSH Terms: conditions — Dyspepsia | interventions — palmidrol

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEA + participant ON-PPI (Active Comparator): Patiënts that on baseline take daily PPI treatment are randomized in the ON-PPI PEA arm or ON-PPI placebo arm
  Interventions: Dietary Supplement: Palmitoylethanolamide
- Placebo + Participant ON-PPI (Placebo Comparator): Patiënts that on baseline take daily PPI treatment are randomized in the ON-PPI PEA arm or ON-PPI placebo arm
  Interventions: Dietary Supplement: Palmitoylethanolamide
- PEA + participant OFF-PPI (Active Comparator): Patiënts that do not take PPI at baseline are randomized in the OFF-PPI PEA arm or OFF-PPI placebo arm
  Interventions: Dietary Supplement: Palmitoylethanolamide
- Placebo + participant OFF-PPI (Placebo Comparator): Patiënts that do not take PPI at baseline are randomized in the OFF-PPI PEA arm or OFF-PPI placebo arm
  Interventions: Dietary Supplement: Palmitoylethanolamide

INTERVENTIONS:
Dietary Supplement: Palmitoylethanolamide — 8-week treatment 3x400 mg per day

SUMMARY:
The goal of this placebo controlled randomized double blind interventional study is to assess the effect of palmitoylethanolamide supplementation in patients with functional dyspepsia The main questions it aims to answer are:

* The efficacy of PEA on functional dyspepsia symptoms measured using the LPDS questionnaire
* The effect of PEA on duodenal mucosal permeability.

Participants will receive an 8-week during treatment with PEA 3x400 mg per day or placebo 3 times per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with functional dyspepsia as diagnosed by the Rome IV criteria.
* Subjects must provide witnessed written informed consent prior to any study procedures being performed.
* Subjects aged 18-70 years old.
* Male or female subjects.
* Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements.
* Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Highly effective birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.

Exclusion Criteria:

* Presence of a history of gastrointestinal surgery other than appendectomy and cholecystectomy.
* Organic gastro-intestinal disease
* Major psychiatric disorder such as major depression
* Presence of coeliac disease, lupus, scleroderma and other systemic auto-immune disease.
* Patients with eosinophilic esophagitis
* Presence of diabetes mellitus
* Active H. Pylori infection or < 6 months after eradication
* Predominant IBS (based on the Rome IV questionnaire)
* Predominant GERD (based on the Rome IV questionnaire)
* Patients taking prohibited medication
* Females who are pregnant or lactating
* Patients not capable to understand or be compliant with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect (change) on the Leuven-postprandial distress scale (LPDS) (0-15), higher score indicating more symptoms) | Comparison after 8 weeks of treatment with placebo or PEA
  Validated questionnaire for measurement of dyspeptic symptoms in functional dyspepsia

SECONDARY OUTCOMES:
Effect of PEA supplementation on duodenal permeability | Comparison after 8 weeks of treatment with placebo or PEA
  Duodenal biopsies in Ussing chambers (measurement of mucosal permeability)
Effect of PEA supplementation on duodenal inflammation | Comparison after 8 weeks of treatment with placebo or PEA
  Counting of mast-cells and eosinophils
Effect of PEA on gastric emptying | Comparison after 8 weeks of treatment with placebo or PEA
  Assessed by gastric emptying breath test

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarnelli G, Pesce M, Seguella L, Lu J, Efficie E, Tack J, Elisa De Palma FD, D'Alessandro A, Esposito G. Impaired Duodenal Palmitoylethanolamide Release Underlies Acid-Induced Mast Cell Activation in Functional Dyspepsia. Cell Mol Gastroenterol Hepatol. 2021;11(3):841-855. doi: 10.1016/j.jcmgh.2020.10.001. Epub 2020 Oct 14. PMID 33065341